CLINICAL TRIAL: NCT00049998
Title: An Open-Label, Multicentre, Randomised, Phase III Study Comparing Oral Topotecan to Intravenous Docetaxel in Patients With Pretreated Advanced Non Small Cell Lung Cancer
Brief Title: Oral Topotecan Versus Intravenous Docetaxel In Pretreated, Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104864-A/387
Record Dates: First submitted 2002-11-18; First posted 2002-11-20 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Nonsmall Cell Lung cancer; advanced; Second-line; topotecan; Hycamtin; oral; docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Topotecan

INTERVENTIONS:
Drug: topotecan

SUMMARY:
The purpose of this study is to collect information on how effective and how well tolerated an oral investigational drug is compared to a standard intravenous drug in patients with pretreated, advanced non-small lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients with advanced non-small cell lung cancer (NSCLC).
* Patients who have received one previous chemotherapy for NSCLC.
* Full recovery from previous chemotherapy.
* Presence of either measurable or non-measurable disease by radiologic study or physical examination.
* At least 3 weeks since last major surgery (a lesser period is acceptable if deemed in the best interest of the patient).
* At least 24 hours since prior radiotherapy providing that marked bone marrow suppression is NOT expected. Patients who have received radiotherapy must have recovered from any reversible side effects (e.g. nausea and vomiting).
* Laboratory criteria: Patients must have adequate bone marrow reserve and adequate kidney and liver function.

Exclusion Criteria:

* Symptoms of brain metastasis (cancer spreading to the brain), requiring treatment with steroids.
* Active infection.
* Severe medical problems other than the diagnosis of NSCLC, that would limit the ability of the patient to follow study guidelines or expose the patient to extreme risk.
* Ongoing or planned chemotherapy, immunotherapy, radiotherapy, or investigational therapy for the treatment of NSCLC.
* Use of investigational drug within 30 days prior to the first dose of study medication.
* Women who are pregnant or lactating.
* Patients of child-bearing potential refusing to practice adequate birth control methods.
* Patients with conditions which might alter absorption of an oral drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760
Dates: Start 2001-10; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
One-year survival rate

SECONDARY OUTCOMES:
overall survival, time to progression, response rate, response duration, time to response, improvement in quality of life and patient well-being, and qualitative and quantitative toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (107):
- Australia (4):
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Ringwood East, Victoria
- Austria (3):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Sankt Pölten
  - GSK Investigational Site, Vienna
- Belgium (4):
  - GSK Investigational Site, Braasschaat
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Liège
- Canada (7):
  - GSK Investigational Site, Sydney, Nova Scotia
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- China (5):
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wangfujing, Beijing
- Czechia (3):
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Kladno
  - GSK Investigational Site, Prague
- Denmark (2):
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Odense C
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Turku
- France (5):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulon Naval
  - GSK Investigational Site, Vesoul
- Germany (8):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Treuenbrietzen, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Berka, Thuringia
- Greece (5):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Papagos, Athens
  - GSK Investigational Site, Rio, Patras
  - GSK Investigational Site, Thessaloniki
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Csorna
  - GSK Investigational Site, Miskolc
- Israel (4):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
- Italy (5):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Verona, Veneto
- GSK Investigational Site, Riga, Latvia
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- Netherlands (5):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Delft
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Leeuwarden
- GSK Investigational Site, Newtown, Wellington, New Zealand
- GSK Investigational Site, Quezon City, Philippines
- Poland (2):
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Portugal (2):
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
- GSK Investigational Site, Singapore, Singapore
- South Africa (3):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Cape Town, Western Province
  - GSK Investigational Site, Port Elizabeth
- Spain (9):
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, La Laguna (Santa Cruz de Tenerife)
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Zurich, Switzerland
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan County
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- Turkey (Türkiye) (2):
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir
- Ukraine (3):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Luhansk
  - GSK Investigational Site, Lviv
- United Kingdom (6):
  - GSK Investigational Site, Dundee, Forfarshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, London, London
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Guildford, Surrey